CLINICAL TRIAL: NCT01881438
Title: Oral Fluoroquinolones and the Risk of Retinal Detachment
Brief Title: An Observational Study of Oral Fluoroquinolones and the Risk of Retinal Detachment
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100940; RRA-7875 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Retinal Detachment
Keywords: Retinal Detachment; Fluoroquinolones; Ciprofloxacin; Levofloxacin; Gatifloxacin; Gemifloxacin; Moxifloxacin; Norfloxacin; Ofloxacin; Beta-Lactam
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants exposed to oral fluoroquinolones: Oral fluoroquinolones in this study are ciprofloxacin, levofloxacin, gatifloxacin, gemifloxacin, moxifloxacin, norfloxacin, and ofloxacin.

SUMMARY:
The purpose of this study is to assess the association of retinal detachment (separation of the retina [the innermost layer of the eyeball] from its connection at the back of the eye) with exposure to oral ciprofloxacin or oral fluoroquinolones.

DETAILED DESCRIPTION:
This is an observational (in which the investigators observe the outcomes of the study participants but do not intervene by, e.g, assigning the treatments) and retrospective (a study in which the exposures and outcomes occurred before the study began) study. It will use data from the Optuminsight and Truven Commercial Claims and Encounters databases, each of which will be evaluated separately using 3 designs: (1) Case-control (a design that compares the cases [study participants], ie, those with retinal detachment to controls, ie, a sample of similar people who did not have a retinal detachment) to assess whether their exposures to fluoroquinolones (FQs) differed. Two case-control studies are planned, one (replication) that mimics a previously reported study, the other (revised) that addresses more potential confounders than did that study , (2) Cohort (a design that follows the participants exposed to FQs and those not exposed to FQs to assess whether the two groups had different risks of developing retinal detachment), (3) Case-only (a design where the exposure history of individuals who had retinal detachment are examined to assess whether they were more likely to have had it when they were exposed to FQs than when they were not).

ELIGIBILITY:
Inclusion criteria:

* At least 1 year of enrollment in the study for medical and pharmacy benefits after their cohort (group) entry (the day of their first ophthalmologist visit) for case-control design
* Oral fluoroquinolone like levofloxacin or ciprofloxacin must be dispensed to participants for cohort design
* At least one visit to an ophthalmologist and enrolled at least for 1 year in the study for medical and pharmacy benefits prior to the date of first occurrence of the exposure of levofloxacin or ciprofloxacin for cohort design
* At least one visit to an ophthalmologist and enrolled at least for 1 year in the study for medical and pharmacy benefits prior to the diagnosis of their first retinal detachment (separation of the retina [the innermost layer of the eyeball] from its connection at the back of the eye) for case-only design

Exclusion criteria:

- Prior diagnosis of retinal detachment , prior diagnosis or procedure for inflammatory conditions of the eyeball, or hospital admission between cohort entry and the date of the retinal detachment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with exposure to oral fluoroquinolones
Sampling Method: Non-Probability Sample
Enrollment: 119924 (Actual)
Dates: Start 2000-01; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of Retinal Detachments With Exposure to Oral Ciprofloxacin or to Oral Fluoroquinolones | 11 years
  Oral fluoroquinolones in this study are gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, and ofloxacin.

SECONDARY OUTCOMES:
Number of Retinal Detachments With Exposure to Oral Ciprofloxacin or to Oral Fluoroquinolones (Revised Case-Control Design) | 11 years
  Oral fluoroquinolones in this study are gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, and ofloxacin. Revised Case-control design is used for assessment of this outcome measure.
Number of Retinal Detachments With Exposure to Individual Oral Fluoroquinolones (Revised Case-Control Design) | 11 years
  Oral fluoroquinolones in this study are gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, and ofloxacin. Revised Case-control design is used for assessment of this outcome measure.
Number of Retinal Detachments With Exposure to Oral Fluoroquinolones Along With Oral Beta-Lactam antibiotic (Case-Control Design) | 11 years
  Oral fluoroquinolones in this study are gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, and ofloxacin. Case-control design is used for assessment of this outcome measure.
Number of Retinal Detachments With Exposure to Oral Levofloxacin and Ciprofloxacin (Cohort Design) | 11 years
  Cohort design is used for assessment of this outcome measure.
Number of Retinal Detachments During the Period of Exposure With Oral Levofloxacin and Ciprofloxacin (Case-Only Design) | 11 years
  Case-only design is used for assessment of this outcome measure.
Number of Retinal Detachments During the Period of non-Exposure to Oral Levofloxacin and Ciprofloxacin (Case-Only Design) | 11 years
  Case-only design is used for assessment of this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC